CLINICAL TRIAL: NCT04127422
Title: Risk Factors for Benign Breast Disease in Young Adult Women. Case-control Study
Brief Title: Risk Factors for Benign Breast Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Professor of Surgery, Mansoura University
Other Study IDs: R.19.08.579
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Benign Breast Disease
Keywords: Benign breast disease; Fibrocystic disease
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients presenting with current symptoms related to the breast. Adult females aged 18-39 years presenting to the breast outpatient clinic with either mastalgia, nodularity and/or discharge.
  A questionnaire, physical examination and bilateral breast ultrasonography will be obtained for all patients.
  A- The questionnaire will contain the following items:
  1. symptoms related to the breast.
  2. other medical history.
  3. menstrual history.
  4. obstetric history.
  5. rapid screener for beverages and fast food consumption.
  6. rapid screener for vegetables and fruit consumption.
  B- Physical examination will specifically records the following:
  1. breast tender point(s).
  2. breast nodularity.
  3. nipple discharge.
  4. weight, height, body mass index (BMI).
  C- bilateral breast ultrasonography for all patients.
  D- breast biopsy when clinically indicated as per hospital policy.
- Control group: Age-matched healthy volunteers with no current medical conditions. Adult females aged 18-39 years with no current breast problems. These healthy volunteers will be asked to complete the same questionnaire as per the Study group and have anthropometric measure.
  A- The questionnaire will contain the following items:
  1. other medical history.
  2. menstrual history.
  3. obstetric history.
  4. rapid screener for beverages and fast food consumption.
  5. rapid screener for vegetables and fruit consumption.
  B- Physical examination will specifically records the following:
  1- weight, height, body mass index (BMI).

SUMMARY:
Benign diseases of the breast are common clinical conditions that affect young women. Complaints related to the breast often cause significant discomfort and mental stress. The following study will try to identify the risk factors that may be associated with symptomatic benign breast diseases. Identification of such factors may help preventing and / or treating these conditions.

DETAILED DESCRIPTION:
Benign breast disease (BBD) is a common cause of hospital visit. In young adults, benign breast conditions surpass cancer as a cause of symptoms related to the breast. However, breast symptoms may be associated with significant distress and may impose diagnostic difficulties. Moreover, certain pathological entities of benign breast conditions are well known to increase the risk of breast cancer.

Identification of modifiable risk factors associated with symptomatic breast disorders has several potential benefits. Modification of such factors may help decrease patients' distress, hospital visits and indirectly decrease the risk of cancer.

the available data point to the possible association of several environmental factors with symptomatic BBD. Most of the available information points to an association of BBD with anthropometric features, growth pattern, family history of breast conditions and dietary consumption. Substantial evidence are however lacking and further studies are strongly required to better characterize the risk factors of the condition.

In this study, the investigators will systematically collect epidemiological, developmental and clinical data in young patients presenting with breast complaints. The association with disease incidence, pattern and histology will be examined.

ELIGIBILITY:
Inclusion Criteria:

* adult females with current symptoms related to the breast.

Exclusion Criteria:

* Current or past malignancy of the breast.
* Discrete breast mass that necessitate work-up to exclude cancer.
* Current psychiatric morbidity.
* Persons unwilling to participate.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult females presenting to the breast outpatient clinic at Mansoura University Oncology Center.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Relative risk of benign breast disease associated with obesity. | This outcome will be assessed at baseline (the first hospital visit).
  For the study and control groups, body mass index will be calculated as the weight (Kg) to square height (m) ratio.
Relative risk of benign breast disease associated with soda beverage consumption. | This outcome will be assessed at baseline (the first hospital visit).
  for the study and control groups, the participant will be asked about soda beverage consumption in the last 30 days. never consumed is scored 0 (lowest score). Three or more times a day is scored 9 (highest score).
Relative risk of benign breast disease associated with caffeine beverages consumption. | This outcome will be assessed at baseline (the first hospital visit).
  for the study and control groups, the participant will be asked about caffeine beverage consumption in the last 30 days. never consumed is scored 0 (lowest score). Three or more times a day is scored 9 (highest score).
Relative risk of benign breast disease associated with parity. | This outcome will be assessed at baseline (the first hospital visit).
  for the study and control groups, the participant will be asked about her parity. response will be either nullipara, primipara, multipara or grand multipara ( 5 or more births).

OTHER OUTCOMES:
Relative risk of benign breast disease associated with hormonal contraception. | This outcome will be assessed at baseline (the first hospital visit).
  for the study and control group, the participant will be asked about current hormonal contraception use.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Cancer center, Al Mansurah, Egypt